CLINICAL TRIAL: NCT00217802
Title: The Effect of Self-regulatory Education on Women With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 289; R01HL060884 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: six-session telephone counseling program

SUMMARY:
The project evaluates an innovative educational intervention using telephone counseling based on self-regulation theory designed to address a problem heretofore overlooked in asthma self-management education: the unique needs of adult female patients.

DETAILED DESCRIPTION:
BACKGROUND:

More than half of the adults with asthma in the US are female. Prevalence of asthma in women appears to be increasing, and morbidity and mortality rates for this group are significantly higher than rates for men. Recent studies point to unique features in women's management of asthma potentially attributable to gender. These include, for example, factors associated with hormonal cycles, (e.g. menses, pregnancy, menopause) and social roles (e.g. household tasks exposing one to environmental triggers, caregiving to children and relatives interfering with asthma management etc.) To date, no rigorously evaluated intervention expressly designed for women with asthma has been reported in the literature.

DESIGN NARRATIVE:

This study is to assess the effectiveness of a gender-specific telephone counseling, self-regulation intervention for women with asthma. To test our hypothesis we employed a randomized controlled design utilizing an intervention group and a control group. The primary outcomes are gender-related asthma management problems, health care utilization, days having symptoms, self-regulation level, management skill, and quality of life. We measure at three time points: baseline before randomization; follow-up I, one year subsequent to randomization; and follow-up II, one year subsequent to follow-up.

ELIGIBILITY:
The study participants are a noninstitutionalized ambulatory sample of women who are willing to participate in the project and meet the following criteria:

1. 18 years of age or older,
2. a diagnosis of asthma,
3. presence of active symptoms,
4. enrolled as a patient in one of the University of Michigan Medical Center asthma-related clinics,
5. listed as having received face-to-face instructions by clinic personnel on peak flow monitoring and proper use of medicine and delivery devices, and
6. not pregnant.

Women who are found to have extenuating circumstances that would prevent them from fully benefiting from the program (e.g., mental illness or terminal illness) are excluded.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Clark — University of Michigan